CLINICAL TRIAL: NCT01740804
Title: A Prospective Observational Study on the Dynamic Changes of CTC Enumeration in Advanced NSCLC With 1st Line Chemotherapy
Brief Title: Dynamic Circulating Tumor Cell (CTC) Changes During the Chemotherapy in NSCLC
Acronym: POLICE
Status: Completed | Type: Observational
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Other Study IDs: CTONG1202
Record Dates: First submitted 2012-11-27; First posted 2012-12-04 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2015-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Cell, Circulating Tumor
Keywords: Circulating tumor cell; Non-small cell lung cancer; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The DNA sample will be rtetained for molecular analysis such as EGFR, KRAS, etc.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Primary endpoint To observe the dynamic changes of CTC during the process of platinum based chemotherapy in advanced NSCLC.

To study the relationship between CTC count and clinical outcome of chemotherapy (ORR and PFS).

Secondary endpoint To study the relationship between CTC and overall survival. To study the molecular feature of CTC, such as epidermal growth factor receptor (EGFR), KRAS, CD117, etc.

DETAILED DESCRIPTION:
This is a prospective observational non-intervention study evaluating the dynamic CTC count during the chemotherapy. Patients provide written informed consent and pass the screening. Peripheral blood will be drawn before and after the first line chemotherapy. Analyze the relationship between CTC count and clinical outcome. The time points of blood drawing are set as following: once prior to 1st cycle of chemotherapy, once 1 week prior to 2nd cycle of chemotherapy, posterior to 4th cycle (or less than 4th cycle) of chemotherapy and once when progressive disease (PD). The specific blood tube CellSave Tube will be used, 7.5ml blood sample every time. One follow-up (including by phone) be made every 3 month after PD until death. The clinical outcome of first line chemotherapy will be ultimately obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically documented, locally advanced or recurrent (stage IIIb and not amenable or combined modality treatment) or metastatic (stage IV) non-small cell lung cancer.
* ECOG performance status of ≤ 2.
* Patients without prior chemotherapy or therapy with systemic anti-neoplastic therapy. Previous adjuvant or neo-adjuvant treatment or combine chemoradiotherapy for stage I to III is permitted if completed > 12 months before enrollment.
* According to routine first line doublet chemotherapy in clinical practice, Cisplatin or carboplatin combined with gemcitabine or paclitaxel or docetaxol or Vinorelbine were recommended.
* Patients must have measurable disease according to the RECIST (version 1.1) criteria.
* Life expectancy of at least 12 weeks.
* Age ≥ 18 years.
* Written (signed) informed Consent to participate in the study.
* Adequate organ function as defined by the following criteria:Liver function: SGOT (AST) and SGPT (ALT) ≤ 2.5 X ULN in the absence of liver metastases or up to 5 X ULN in case of liver metastases. Total bilirubin ≤ 1.5ULN.Bone marrow function: Granulocyte count ≥ 1,500/mm3 and platelet count ≥100,000/mm3 and hemoglobin ≥90g/dl. Renal function: serum creatinine ≤ 1.5 ULN or creatinine clearance ≥ 60 ml/min. (based on modified Cockcroft-Gault formula).
* For all females of childbearing potential a negative serum/urine pregnancy test must be obtained within 48 hours before enrollment. Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential.

Exclusion Criteria:

* Patients with prior chemotherapy or therapy with systemic anti-cancer therapy including target therapy. Previous adjuvant or neo-adjuvant treatment for non-metastatic disease is permitted if completed ≥ 6 months before the enrollments.
* Patients with history of any other malignancies within 5 years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer).
* Patients who have brain metastasis or spinal cord compression. It is permitted if the patient has been treated with surgery and/or radiation with evidence of stable disease for at least 4 weeks.
* Patients who are at risk (in the investigator's opinion) of transmitting human immunodeficiency virus (HIV) through blood or other body fluids.
* Nursing or lactating women.
* Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study.
* Unwilling to write informed consent to participate in the study.
* Patients who is unwilling to accept the follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced NSCLC (stage IIIb/IV or recurrent NSCLC)
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2012-11; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
dynamic CTC changes during chemotherapy | baseline, 3 weeks and up to progression disease of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Long Wu, MD, Principal Investigator — Guangdong General Hospital & Guangdong Academy of Medical Sciences
Locations (1):
- Guangdong general hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Wang Z, Zhang XC, Feng WN, Zhang L, Liu XQ, Guo WB, Deng YM, Zou QF, Yang JJ, Zhou Q, Wang BC, Chen HJ, Tu HY, Yan HH, Wu YL. Circulating tumor cells dynamics during chemotherapy predict survival and response in advanced non-small-cell lung cancer patients. Ther Adv Med Oncol. 2023 Apr 22;15:17588359231167818. doi: 10.1177/17588359231167818. eCollection 2023. PMID 37113733